CLINICAL TRIAL: NCT05247905
Title: Phase II Randomized, Prospective Trial of Lutetium Lu 177 Dotatate PRRT Versus Capecitabine and Temozolomide in Well-Differentiated Pancreatic Neuroendocrine Tumors
Brief Title: Comparing Capecitabine and Temozolomide in Combination to Lutetium Lu 177 Dotatate in Patients With Advanced Pancreatic Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A022001; NCI-2021-14404 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Pancreatic Neuroendocrine Tumor; Unresectable Pancreatic Neuroendocrine Carcinoma
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — lutetium Lu 177 dotatate; Capecitabine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (lutetium Lu 177 dotatate) (Experimental): Patients receive lutetium Lu 177 dotatate IV over 30 minutes on day 1. Treatment repeats every 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lutetium Lu 177 Dotatate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (capecitabin, temozolomide) (Experimental): Patients receive capecitabine PO BID days 1-14 and temozolomide PO QD on days 10-14. Treatment repeats every 4 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Temozolomide; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Lutetium Lu 177 Dotatate — Given IV
  Arms: Arm I (lutetium Lu 177 dotatate)
Drug: Capecitabine — Given PO
  Arms: Arm II (capecitabin, temozolomide)
Drug: Temozolomide — Given PO
  Arms: Arm II (capecitabin, temozolomide)
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm I (lutetium Lu 177 dotatate)

SUMMARY:
This phase II trial compares capecitabine and temozolomide to lutetium Lu 177 dotatate for the treatment of pancreatic neuroendocrine tumors that have spread to other parts of the body (advanced) or are not able to be removed by surgery (unresectable). Chemotherapy drugs, such as capecitabine and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radioactive drugs, such as lutetium Lu 177 dotatate, may carry radiation directly to tumor cells and may reduce harm to normal cells. The purpose of this study is to find out whether capecitabine and temozolomide or lutetium Lu 177 dotatate may kill more tumor cells in patients with advanced pancreatic neuroendocrine tumors.

DETAILED DESCRIPTION:
This phase II trial compares capecitabine and temozolomide to lutetium Lu 177 dotatate for the treatment of pancreatic neuroendocrine tumors that have spread to other parts of the body (advanced) or are not able to be removed by surgery (unresectable). Chemotherapy drugs, such as capecitabine and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radioactive drugs, such as lutetium Lu 177 dotatate, may carry radiation directly to tumor cells and may reduce harm to normal cells. The purpose of this study is to find out whether capecitabine and temozolomide or lutetium Lu 177 dotatate may kill more tumor cells in patients with advanced pancreatic neuroendocrine tumors.

The primary and secondary objectives of the study:

PRIMARY OBJECTIVE:

I. To determine the differences in median progression-free survival (PFS) for lutetium Lu 177 dotatate peptide receptor radionuclide therapy (PRRT) when compared to capecitabine and temozolomide (CAPTEM) in patients with locally advanced or metastatic progressive, well-differentiated pancreatic neuroendocrine tumors (pNETs).

SECONDARY OBJECTIVES:

I. To evaluate and compare the overall survival (OS) of patients receiving lutetium Lu 177 dotatate versus (vs.) CAPTEM.

II. To evaluate and compare time to response, time to maximum response, and overall response rates (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 between both arms.

III. To evaluate and compare duration of response and time to progression among both arms.

IV. To evaluate and compare treatment related toxicities between the arms. V. To compare global health status/quality of life as measured with the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30 from baseline through 18 months between patients with pNET treated with lutetium Lu 177 dotatate PRRT versus capecitabine and temozolomide.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive lutetium Lu 177 dotatate intravenously (IV) over 30 minutes on day 1. Treatment repeats every 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive capecitabine orally (PO) twice daily (BID) days 1-14 and temozolomide PO once daily (QD) on days 10-14. Treatment repeats every 4 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or pathologic documentation: well-differentiated pancreatic neuroendocrine tumor (G1, G2, or well-differentiated G3) confirmed by local histology and/or pathology
* Functional or nonfunctional tumors are allowed
* Stage: locally unresectable or metastatic disease
* Tumor Site: neuroendocrine tumor of pancreatic primary site
* Radiologic evaluation: tumor must have shown somatostatin receptor (SSTR) positivity on 68Ga-DOTATATE PET or other SSTR-PET scan in the 12 months prior to registration; however, documentation of SSTR positivity in the 6 months prior to registration is preferred. SSTR positivity is defined as uptake greater than background liver in all measurable lesions
* Patients are eligible if they meet one of the following criteria:

  * Previously untreated patients with grade 2 or 3 disease AND with symptoms of either disease bulk causing pain, anorexia, early satiety, large effusions/ascites, abdominal pain, abdominal fullness due to hepatomegaly, dyspnea) OR incompletely controlled symptoms of hormone excess despite somatostatin analogue (SSA) and supportive care (including but not limited to: diarrhea, hypercalcemia, hypoglycemia, hyperglycemia, flushing, Cushing's syndrome). Patient may have been started on SSA for up to 2 months for attempted symptom control without disease progression prior to registration
  * Patients previously treated with SSA only and with disease progression by RECIST in prior 12 months
  * Patients previously treated with SSA and one or more prior systemic therapy must have received prior anti-vascular endothelial growth factor (VEGF) pathway therapy inhibitor OR have contraindication to anti-VEGF therapy (including but not limited to: uncontrolled hypertension [systolic blood pressure [SBP] > 150 and/or diastolic blood pressure [DBP] > 90 despite medical management], stage IIB or greater heart disease, angina pectoris, prior arterial [ATE] and venous thromboembolic [VTE] events in the past 6 months, gastrointestinal [GI] bleed in the last 6 months) and disease progression by RECIST in prior 12 months
  * Patients previously treated with more than 2 lines of therapy, not including anti VEGF therapy, but with NET related symptoms as outlined in first bullet (pain, anorexia, early satiety, large effusions/ascites, abdominal pain, abdominal fullness due to hepatomegaly, anorexia, early satiety, dyspnea) OR incompletely controlled symptoms of hormone excess despite somatostatin analogue (SSA) and supportive care (including but not limited to: diarrhea, hypercalcemia, hypoglycemia, hyperglycemia, flushing, Cushing's syndrome).
  * Any patient with disease progression by RECIST criteria in < 4 months
* Patients must have measurable disease per RECIST v1.1 by computer tomography (CT) scan or magnetic imaging (MRI). Any lesions which have undergone percutaneous therapies or radiotherapy after starting protocol therapy should not be considered measurable unless the lesion has clearly progressed since the procedure.

  * Lesions must be accurately measured in at least one dimension (longest diameter to be recorded) as >= 1 cm with CT or MRI (or shortest diameter >= 1.5 cm for lymph nodes). Non-measurable disease includes disease smaller than these dimensions or lesions considered truly non- measurable including: leptomeningeal disease, bone metastases, ascites, pleural or pericardial effusion, lymphangitic involvement of skin or lung.
* Prior treatment with tyrosine kinase inhibitors (TKIs) such as mammalian target of rapamycin (mTOR) inhibitors (e.g. everolimus, temsirolimus, etc.) or VEGF pathway inhibitors (e.g. sunitinib, pazopanib, cabozantinib, bevacizumab, etc.) are allowed
* Prior treatment with hepatic intra-arterial embolic therapies is allowed if there is recovery from all toxicities, measurable lesions do not include embolized liver unless there has been clear subsequent progression, all measurable lesions are somatostatin receptor avid, and treatment completed at least 2 months prior to registration
* Prior treatment with cryoablation or thermal/radiofrequency ablation of metastases is allowed if there is recovery from all toxicities, measurable lesions do not include treated metastases, and treatment completed at least 2 months prior to registration
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Creatinine =< 1.5 x upper limit of normal (ULN) OR calculated (calc.) creatinine clearance >= 30 mL/min (calculated by the Cockcroft-Gault equation)
* Total bilirubin =< 1.5 x ULN (in patients with liver metastases or known Gilbert's syndrome, total bilirubin must be =< 3.0 x ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x ULN
* Albumin >= 3.0 g/dL
* Concurrent somatostatin analog use while on protocol therapy is allowed provided that the patient:

  * Has a functional tumor (evidence of peptide hormones and/or bioactive substances associated with a clinical hormone syndrome such as carcinoid syndrome or Cushing's syndrome)
  * Has been on a stable dose of somatostatin analog therapy for at least three months
  * Has previously demonstrated radiographic disease progression while on somatostatin analog therapy. For subjects receiving lutetium Lu 177 dotatate, there should be a minimum of 14 days between long-acting somatostatin analogue and lutetium Lu 177 dotatate dosing. Short-acting somatostatin analogs should not be administered within 24 hours of lutetium Lu 177 dotatate dosing. Following lutetium Lu 177 dotatate dosing, long-acting somatostatin analogs may be administered between 4 and 24 hours after each dose

Exclusion Criteria:

* Patients with poorly differentiated neuroendocrine carcinoma (large cell histology or small cell histology) are not eligible
* No prior temozolomide, dacarbazine, capecitabine, 5-FU, or any PRRT for treatment of the pNET
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects

  * Therefore, for women of childbearing potential only, a negative pregnancy test done =< 14 days prior to registration is required
* No known brain metastases unless adequately treated, demonstrated to be stable, and off all treatment (including steroids) for at least 2 months prior to registration
* No uncontrolled congestive heart failure (New York Heart Association [NYHA] II, III, IV).
* No significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may pose a risk to patient safety
* No "currently active" second malignancy other than non-melanoma skin cancers or cervical carcinoma in situ. Patients are not considered to have a "currently active" malignancy if they have completed therapy or are on adjuvant hormonal therapy and are free of disease for >= 3 years
* No known medical condition causing an inability to swallow and no known impairment of gastrointestinal function that may significantly alter the absorption of an oral agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2033-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 8 years from randomization
  Progression free survival (PFS) will be compared between the two treatment arms using Kaplan-Meier methods. The hazard ratio (HR) and median PFSwill be estimated along with corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) at 2 years | At 2 years from randomization
  Kaplan-Meier methodology will be used to estimate the PFS rate at 2 years.
Progression Free Survival (PFS) at 3 years | At 3 years from randomization
  Kaplan-Meier methodology will be used to estimate the PFS rate at 3 years.
Time to progression (TTP) | Up to 8 years from randomization
  Kaplan-Meier methodology will be used to estimate the median time to progression (TTP).
Overall survival (OS) | Up to 8 years from study registration
  Kaplan-Meier methodology will be used to estimate the median overall survival (OS). OS is defined as randomization to the time of death due to any cause (or censored at the time of last contact for surviving patients and those lost to follow-up).
Objective response rate (ORR) | Up to 8 years from randomization
  The response rate (percentage) is the percent of patients whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST 1.1 criteria. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients. Response rates (including complete and partial response) will be tested using Fisher's exact test.
Time-to response | Up to 8 years from randomization
  Kaplan-Meier methodology will be used to estimate the median time-to-response. Time-to-response will be defined as the time from randomization to the first tumor response, for those patients having achieved an objective response.
Duration of response | Up to 8 years from randomization
  Kaplan-Meier methodology will be used to estimate the median duration of response. Duration of response will be defined as the time from first assessment with documented response (PR or CR) to the time of progression and/or death. Patients who are still responding as of their last evaluation will be censored at the time point. If we observed documented deaths without progression, we will further evaluate this endpoint with death without progression treated as a competing risk.
Incidence of adverse events | Up to 8 years from randomization
  Patients will be evaluated for adverse events using the National Cancer Institute Common Toxicity Criteria for Adverse Events version 5.0. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported.
Change in Overall Health Question (Q29) from the EORTC QLQ-C30 questionnaire | At baseline up to 18 months
  To evaluate between-arm differences in patient-reported global health status from baseline through 18 months, the area under the curve will be calculated as a summary statistic for each arm based on estimates from a mixed model for patient-reported global health status/quality of life as assessed by the EORTC QLQ-C30 at baseline, 3, 6, 12, and 18 months.
Change in Overall Quality of Life Question (Q30) from the EORTC QLQ-C30 questionnaire | At baseline up to 18 months
  To evaluate between-arm differences in patient-reported quality of life from baseline through 18 months, the area under the curve will be calculated as a summary statistic for each arm based on estimates from a mixed model for patient-reported global health status/quality of life as assessed by the EORTC QLQ-C30 at baseline, 3, 6, 12, and 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J. b, MD, Study Chair — Mayo Clinic
Locations (171):
- United States (171):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Bay Area Tumor Institute, Oakland, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Outpatient Center - Oak Lawn, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Mercy Health - Paducah Cancer Center, Paducah, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Mount Sinai Hospital, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Jefferson Healthcare, Port Townsend, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Health Center - Greenfield, Greenfield, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin